CLINICAL TRIAL: NCT00343447
Title: Phase II Randomized Trial of Early Versus Late Vaccination in Patients With High Risk CLL
Brief Title: Cyclophosphamide and Rituximab Followed By Vaccine Therapy in Treating Patients With Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0579 CDR0000481362; P30CA006973 (NIH); JHOC-J0579; JHOC-NA_00000982
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — FANG vaccine; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: autologous tumor cell vaccine
Biological: rituximab
Drug: cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Vaccines may help the body build an effective immune response to kill cancer cells. Giving cyclophosphamide and rituximab together with vaccine therapy may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying cyclophosphamide and rituximab followed by two different schedules of vaccine therapy to compare how well they work in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and toxicity of cyclophosphamide and rituximab in patients with previously untreated, high-risk chronic lymphocytic leukemia.
* Determine, preliminarily, the efficacy and toxicity of early vs delayed administration of vaccine therapy comprising KGEL and autologous tumor cells after cyclophosphamide and rituximab in these patients.
* Compare the magnitude of the T-cell response to early vs delayed administration of this vaccine after rituximab and cyclophosphamide and correlate these responses with the extent of immune reconstruction.

OUTLINE: This is a randomized phase II study for patients with asymptomatic or minimally symptomatic, untreated CLL with poor-risk features.

Patients undergo peripheral blood collection for vaccine production. Patients then receive rituximab IV over at least 4 hours on days 1 and 2 in course 1 and on day 1 only in subsequent courses and cyclophosphamide IV over 1 hour on day 1. Treatment with rituximab and cyclophosphamide repeats every 21 days for up to 6 cycles in the absence of disease progression. Patients undergo evaluation 4 weeks after completion of rituximab and cyclophosphamide. Patients achieving partial or complete response are randomized to 1 of 2 vaccine treatment arms.

* Arm I (early administration): Beginning 2 weeks after evaluation, patients receive vaccine therapy comprising an autologous tumor admixed with an allogeneic vaccine (KGEL) that produces sargramostim (GM-CSF) and autologous tumor cells intradermally. Treatment repeats every 3 weeks for 6 courses in the absence of unacceptable toxicity.
* Arm II (late administration): Beginning 20 weeks after evaluation, patients receive vaccine therapy comprising KGEL and autologous tumor cells intradermally. Treatment repeats every 3 weeks for 6 courses in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL)
* Meets 1 of the following high-risk features:

  * 17p deletion by fluorescent in situ hybridization (FISH)
  * 11q deletion by FISH
  * Unmutated immunoglobulin heavy chain variable region (IgVH) genes, defined as ≥ 98% homology with germline in a Clinical Laboratory Improvement Act (CLIA) approved laboratory
* Any stage disease
* Previously untreated disease

  * Not requiring immediate treatment
* Absolute lymphocyte count ≥ 20,000/mm³

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2 mg/dL (unless secondary to obstructive cholestasis from lymphadenopathy or Gilbert's disease)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infections requiring oral or intravenous antibiotics
* No autoimmune disorder (e.g., autoimmune hemolytic anemia) requiring corticosteroids before the start of study vaccination
* No other malignancy except nonbasal cell skin cancer, carcinoma in situ of the cervix, or tumor that was treated with curative intent ≥ 2 years ago

PRIOR CONCURRENT THERAPY:

* No prior therapy for CLL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Efficacy and toxicity
T-cell response to early versus late vaccine therapy comprising KGEL and autologous tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L. Kasamon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States